CLINICAL TRIAL: NCT03293004
Title: Effects of Hydrolyzed Collagen and Vitamin C on Collagen Synthesis and Explosive Performance
Brief Title: Collagen Vitamin C Dose Response Performance
Acronym: Collagen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1042848
Record Dates: First submitted 2017-09-15; First posted 2017-09-26 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: collagen; tendon; procollagen type I N-terminal; athletes; vitamin C; hydrolyzed collagen
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: A double blinded cross over design where subject are randomized to consume all 5 intervention doses.
Who Masked: Participant, Investigator
Masking Description: All nutritional interventions taste and look similar and are prepared for subjects in opaque bottles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hydrolyzed collagen (Experimental): First, we aim to determine the optimal amount of hydrolyzed collagen with a constant dose of vitamin C in humans to increase a marker of collagen synthesis (PINP). In a randomized, double-blinded, crossover design subjects consume a nutritional supplement with varying doses of hydrolyzed collagen (control (0 g), 5 10, 20 and 30 g hydrolyzed collagen) with a constant dose of vitamin C (50 mg). Each intervention will be separated by a 6-day wash out. Subjects will be asked to consume the supplement 1 hour before 6-min of jump rope exercise. Following completion of exercise, subjects will remain in the lab in a rested state for the subsequent 4 hours. After 4 hours and 24 hours blood samples will be collected. Blood samples will be used for PINP analysis.
  Interventions: Dietary Supplement: Hydrolyzed collagen
- Vitamin C (Experimental): Second, we aim to determine the optimal amount of vitamin C with the determined optimal dose of hydrolyzed collagen in humans to increase a marker of collagen synthesis (PINP). In a randomized, double-blinded, crossover design subjects consume a nutritional supplement with varying doses of vitamin C (0 (control), 50, 250 and 500 mg) with an optimized dose of hydrolyzed collagen as determined from the first arm. Each intervention will be separated by a 6-day wash out. Subjects will be asked to consume the supplement 1 hour before 6-min of jump rope exercise. Following completion of exercise, subjects will remain in the lab in a rested state for the subsequent 4 hours. After 4 hours and 24 hours blood samples will be collected. Blood samples will be used for PINP analysis.
  Interventions: Dietary Supplement: Vitamin C
- Optimized Collagen and Vitamin C supplement (Experimental): The findings from the first 2 arms of the study will be used to inform a training-based study aimed to determine whether exercise together with this optimal dose of hydrolyzed collagen and vitamin C is sufficient to improve rate of force development (RFD) and performance. A gummy food will be developed with the optimized dose of hydrolyzed collagen and vitamin C as well as a placebo. In a randomized, double-blinded, parallel design with subjects undertake a 3 week exercise protocol. The supplement will be ingested 1 hour prior to each exercise session (Monday/Wednesday/Friday). Exercise testing to assess rate of force development (RFD) will take place at the end of each week (Fridays) and these outcomes will be the basis for determining the effects of the nutrition intervention on performance.
  Interventions: Dietary Supplement: Optimized Hydrolyzed Collagen and Vitamin C
- Gummy Placebo (Placebo Comparator): A gummy food will be developed with the optimized dose of hydrolyzed collagen and vitamin C as well as a placebo. In a randomized, double-blinded, parallel design with subjects undertake a 3 week exercise protocol. The supplement or placebo will be ingested 1 hour prior to each exercise session (Monday/Wednesday/Friday). Exercise testing to assess rate of force development (RFD) will take place at the end of each week (Fridays) and these outcomes will be the basis for determining the effects of the nutrition intervention on performance.
  Interventions: Dietary Supplement: Gummy Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolyzed collagen — Escalating dose of Hydrolyzed collagen
  Arms: Hydrolyzed collagen
Dietary Supplement: Vitamin C — Escalating dose of Vitamin C
  Arms: Vitamin C
Dietary Supplement: Optimized Hydrolyzed Collagen and Vitamin C — combination of optimized doses of Hydrolyzed Collagen and Vitamin C
  Arms: Optimized Collagen and Vitamin C supplement
Dietary Supplement: Gummy Placebo — Gummy placebo
  Arms: Gummy Placebo

SUMMARY:
Previous work has shown that gelatin supplementation could increase collagen synthesis in humans. In this study subjects consume placebo, 5 or 15 g of gelatin with a standard amount of vitamin C (48 mg) 1 hour before 6 minutes of jump rope exercise. The feeding and exercise intervention was repeated every 6 hours while the subjects were awake for three days and the amount of the amino terminal procollagen I peptide (PINP) was determined; a marker of collagen synthesis, in the blood. Consistent with the hypothesis that gelatin increases collagen synthesis in humans; the amount of PINP in the 15 g gelatin group was significantly higher than either the placebo or the 5 g groups. These data conclusively demonstrate that gelatin supplementation can increase exercise-induced collagen synthesis in humans. Hydrolyzed collagen has a similar amino acid profile, in particular with high concentrations of glycine, proline, hydroxyproline, and arginine. Thus the current study aims to precisely map out the dose response relationship of hydrolyzed collagen and vitamin C on PINP and to determine the optimal dose to achieve maximal increased in PINP levels.

DETAILED DESCRIPTION:
In preliminary work investigating the physiological determinants of maximal performance in throwing events, researchers found that the best predictor of elite performance was the rate of force development (RFD; Force (N) x time (sec)) when performing and isometric squat. Therefore, it is not surprising that in order to maximize performance, athletes train to optimize RFD.

RFD is determined by three factors:

1. Neural activation of the muscles
2. Type of motor protein (fast or slow myosin)
3. Force transfer Interestingly, performance in power movements (that are highly dependent on RFD) like vertical jump is closely related to tendon stiffness and inversely related to muscle size. This indicates that force transfer, in the form of tendon stiffness, plays an important role in performance and can explain a large amount of variance in determining an athlete's ability to rapidly develop force during a dynamic movement.

The stiffness of a tendon is determined by the amount and cross-linking of collagen within the tissue. Acute exercise is known to increase collagen synthesis as well as the expression of the primary enzyme involved in collagen cross-linking, lysyl oxidase. The result is a denser and stiffer tissue after training. Even though the relationship between exercise and collagen synthesis is known, whether this measure of performance can be improved with nutritional interventions has not been determined.

A recent study looking at amino acid levels following consumption of increasing doses of gelatin (derivative of collagen) in human subjects has shown that the key primary and trace amino acids found in collagen increase in human serum after consuming gelatin. Further, the peak of these amino acids occurs 60 minutes after consuming the gelatin supplement. Therefore, consuming a collagen supplement 1 hour before an exercise intervention should maximize delivery of amino acids to bone and other connective tissues.

To determine whether the gelatin supplement could increase collagen synthesis in humans, subjects consumed placebo, 5 or 15 g of gelatin with a standard amount of vitamin C (48 mg) 1 hour before 6 minutes of jump rope exercise. The feeding and exercise intervention was repeated every 6 hours while the subjects were awake for three days and the amount of the amino terminal procollagen I peptide (PINP) was determined; a marker of collagen synthesis, in the blood. Consistent with the hypothesis that gelatin increases collagen synthesis in humans; the amount of PINP in the 15 g gelatin group was significantly higher than either the placebo or the 5 g groups. These data conclusively demonstrate that gelatin supplementation can increase exercise-induced collagen synthesis in humans.

Similarly, supplementation with collagen hydrolysate has previously been shown to improve cartilage function in a randomized clinical trial in patients with osteoarthritis [9]. McAlindon and colleagues showed that consuming 10 g of collagen hydrolysate per day resulted in an increase in gadolinium enhanced MRI of collagen [9]. This finding suggests that the hydrolyzed collagen increased cartilage formation. In agreement with this finding, a 24-week randomized clinical trial in athletes showed that 10 g of GELITA® collagen hydrolysate significantly decreased knee pain. Mouse studies using C14 labeled hydrolyzed collagen hydrolysate demonstrated that >95% of the hydrolyzed collagen was absorbed in the first 12 hours after feeding. Interestingly, even though tracer from a separate C14 labeled proline could be incorporated into skin collagen at the same rate as tracer from hydrolyzed collagen, tracer from the hydrolyzed collagen was incorporated into the collagen of cartilage and muscle two-fold more than the tracer from proline. These data suggest that musculoskeletal collagen synthesis is greater in response to gelatin or hydrolyzed collagen than to the individual amino acids.

Even though the blood measure of PINP levels likely reflects bone collagen synthesis, using an engineered ligament model, a similar response has been demonstrated in tendons/ligaments treated with serum from people 1 hour after supplementation with gelatin. This work has shown that in the presence of serum isolated from the 5 and 15 grams of gelatin groups a step-wise increase in the collagen content of the ligaments. From this work, it can be ascertained that PINP can be used dependably as an indirect marker of collagen synthesis and that the changes observed in bone (blood levels) reflect what is occurring in other connective tissues as well.

The current study aims to precisely map out the dose response relationship of hydrolyzed collagen and vitamin C on PINP and to determine the optimal dose to achieve maximal increased in PINP levels. Secondly, whether this optimal dose of hydrolyzed collagen and vitamin C, taken before training is sufficient to improve RFD and performance will be determined. To achieve this goal, subjects will first consume increasing doses of hydrolyzed collagen (0 (control), 5, 10, 20 and 30 g) alongside a constant amount of vitamin C (50 mg). Once the optimal dose of hydrolyzed collagen is determined this dose will be administered with increasing doses of vitamin C (0 (control), 50, 250, 500 mg) to determine the optimal dose of vitamin C to maximize PINP levels. Both hydrolyzed collagen and vitamin C supplementation will be given 1 hour before 6 minutes of jump rope exercise.

After the optimal doses of hydrolyzed collagen and vitamin C are determined, the effects of the optimal dose of hydrolyzed collagen and vitamin C on performance will be assessed. Subjects will undergo an explosive/power-based exercise training program three days a week (Monday/Wednesday/Friday) for three weeks. The hydrolyzed collagen and vitamin C will be ingested 1 hour before each training session. Baseline exercise testing will take place at week 0, then exercise testing will occur on Friday of each week (week 1, 2 and 3). Subjects will undergo a series of tests to determine the RFD in the isometric squat, and countermovement and squat jump height.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate level male athletes between 18 - 25 years of age
* Currently registered/participating as an intercollegiate athlete
* < 3 musculoskeletal injuries in the past year
* No health or dietary restriction that would be affected by the supplementation protocol.

Exclusion Criteria:

* History of more than 3 musculoskeletal injuries within the past 12 months.
* Health, dietary restriction or diet that would be affected by the supplementation protocol.
* Then initial phases of this study will be performed in males since collagen synthesis varies significantly throughout the menstrual cycle in females. Since collagen in the main outcome measure for this study this natural variation would confound the initial phase of the work. Provided this work proves successful then we will aim to perform similar studies in females.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
  Then initial phases of this study will be performed in males since collagen synthesis varies significantly throughout the menstrual cycle in females. Since collagen in the main outcome measure for this study this natural variation would confound the initial phase of the work. • Provided this work proves successful then we will aim to perform similar studies in females.
Enrollment: 23 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
PINP Levels | 9 weeks
  To determine optimal dose of supplemental hydrolyzed collagen and vitamin C required to maximally elevate PINP levels (a marker of collagen synthesis) in healthy athletes.
Rate of force development (RFD) | 3 weeks
  a measure of explosive strength

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No